CLINICAL TRIAL: NCT05814094
Title: Red Blood Cell Transfusion in ECMO - A Feasibility Trial
Acronym: ROSETTA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: ANZIC-RC/HB001
Record Dates: First submitted 2022-11-22; First posted 2023-04-14 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Blood Loss Anemia; Extracorporeal Membrane Oxygenation Complication; Disability Physical; Cognitive Ability, General; Functional Status
Keywords: Hb; RBC transfusion; ECMO; feasibility; safety; blood transfusion; Australia; blood products; ICU; critical care; intensive care; bleeding; transfusion; Hb values
MeSH Terms: conditions — Hemorrhage | interventions — Erythrocyte Transfusion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Restrictive Transfusion Trigger Group (Active Comparator): if a patient's Hb concentration reads ≤ 70g/L, one unit of RBC will be transfused. Additional units can be prescribed if required to raise the Hb concentration to above 70g/L.
  Interventions: Other: Red Blood Cell Transfusion
- Liberal Transfusion Trigger Group (Active Comparator): if a patient's Hb concentration reads ≤ 90g/L, one or more units of RBC will be transfused. Additional units can be prescribed to raise the Hb concentration to greater than 90g/L
  Interventions: Other: Red Blood Cell Transfusion

INTERVENTIONS:
Other: Red Blood Cell Transfusion — Following randomisation, if a patient's Hb concentration reads ≤ 70g/L, one unit of RBC will be transfused within 12 hours of the result becoming available. Additional units can be prescribed if required to raise the Hb concentration to above 70g/L. A transfusion above the restrictive threshold of 70g/L is discouraged.
  Arms: Restrictive Transfusion Trigger Group
Other: Red Blood Cell Transfusion — Following randomisation, if a patient's Hb concentration reads ≤ 90g/L, one or more units of RBC will be transfused in order to raise the Hb concentration to greater than 90g/L within 12 hours of the result becoming available. A decision not to transfuse below the threshold of 90g/L is discouraged.
  Arms: Liberal Transfusion Trigger Group

SUMMARY:
Extracorporeal Membrane Oxygenation (ECMO) is an invasive and resource intense treatment used to support critically ill patients who have suffered severe cardiac arrest, cardiac failure or respiratory failure (including severe cases of COVID-19). ECMO acts as a mechanical circulatory support temporarily replacing the function of the heart or lungs by oxygenating blood and removing carbon dioxide, allowing time for these organs to recover. Many critically ill patients, including those on ECMO, have an increased risk of bleeding and reduced production/increased destruction of red blood cells (RBCs). This can lead to anaemia (haemoglobin levels <120 g/l), a condition where the body lacks enough healthy RBCs to carry enough oxygen to the body's tissues. Therefore, patients on ECMO frequently require RBC transfusion, with clinicians having to decide if administering an RBC transfusion (with its associated risks) is higher than tolerating complications of anaemia.

ROSETTA is a feasibility study that aims to determine the safety and feasibility of randomizing patients on ECMO to a restrictive RBC transfusion strategy (maintain Hb concentration above 70g/L) or to a more liberal transfusion strategy (maintain Hb concentration above 90g/L). Feasibility is defined as the ability to achieve a mean separation of at least 10g/L between the average lowest daily haemoglobin values in the two study groups.

DETAILED DESCRIPTION:
A recent Cochrane analysis recommended a transfusion strategy that minimises the use of RBC transfusions in critically ill patients (by tolerating anaemia to avoid the adverse effects of an RBC transfusion). However, the analysis acknowledges that the degree of anaemia which can be tolerated by such patients is unknown, especially in patients suffering from conditions that limit oxygen delivery to the organs (like cardiac disease). As a result, the Australian Blood Authority's guidelines recommend an RBC transfusion to a patient at an Hb concentration of less than 70 g/L, while a transfusion at a Hb between 70 and 90 g/L should be based on the need to relieve clinical signs and symptoms of anaemia. However, this range is broad, and many studies in the general critically ill cohort have shown lower transfusion triggers are non-inferior to higher transfusion triggers.

No studies have been completed directly evaluating transfusion triggers in the ECMO patient cohort. ECMO patients differ to the general critically ill cohort as they have different physiological requirements, are at higher-risk for poor outcomes, and have an increased requirement for transfusions. Hb is a key driver of oxygen delivery (DO2), and critically ill ECMO patients are more commonly exposed to low DO2 due to low cardiac output and borderline oxygenation. Therefore, studies must be done to evaluate the optimal transfusion trigger/s (as determined by Hb concentration) that optimise mortality and long-term outcomes of ECMO patients.

Should the ROSSETTA Pilot results indicate adequate separation of at least 10g/L between the two study groups, and that patient safety has not been adversely affected by the trial methods, feasibility will be deemed confirmed and the protocol not in need of modification prior to full trial commencement. At this point the ROSETTA Pilot will be transitioned into the Red Blood Cell Transfusion Domain, within RECOMMEND Platform Trial. The Primary and Secondary outcomes of the trial at large, will be answered during this stage.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving ECMO
* Age: 18 years or older

Exclusion Criteria:

* Contraindication to RBC transfusion (including known patient preference)
* Limitations of care put in place either through patient wishes or the treating medical teams
* ECMO treatment for more than 12 hours. The start of ECMO is defined as the time of initiation of extracorporeal blood flow unless ECMO was initiated during a surgical intervention in which case the start is defined as the arrival time into the initial ICU.
* The treating physician anticipates that ECMO treatment will cease before the end of tomorrow
* Where the treating physician deems the study is not in the patient's best interest
* Where the treating physician has concern regarding patient ability to tolerate restrictive or liberal transfusion trigger thresholds
* Patients actively listed for a solid organ transplant
* Patients who are suspected or confirmed to be pregnant
* Previous ECMO treatment during the same hospital admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Difference in average lowest daily Hb concentration | From date of randomization to the end of the intervention (assessed up to day 28)
  Primary Outcome Measure

SECONDARY OUTCOMES:
Enrolment Rate | through study completion, an average of 2 years
  Feasibility Outcome
Reasons for not entering eligible patients into the study | through study completion, an average of 2 years
  Feasibility Outcome
Mean pre-transfusion Hb concentration immediately prior to an RBC transfusion | through study completion, an average of 2 years
  Feasibility Outcome
Proportion of RBC transfusions given according to allocated trigger | through study completion, an average of 2 years
  Feasibility Outcome
Time from measured Hb trigger value to transfusion | through study completion, an average of 2 years
  Feasibility Outcome
Number of RBC transfusions given prior to randomization | through study completion, an average of 2 years
  Feasibility Outcome
Frequency for not transfusing a patient who has reached a transfusion trigger | through study completion, an average of 2 years
  Feasibility Outcome
Reason/s for not transfusing a patient who has reached a transfusion trigger | through study completion, an average of 2 years
  Feasibility Outcome
Number of protocol deviations | through study completion, an average of 2 years
  Feasibility Outcome
Number and nature of Serious Adverse Events (SAEs) | through study completion, an average of 2 years
  Safety and effectiveness outcome
Total blood products used | through study completion, an average of 2 years
  Safety and effectiveness outcome
Major bleeding events (defined by ISTH criteria) | through study completion, an average of 2 years
  Safety and effectiveness outcome
Clinically relevant non-major bleeding events: GI haemorrhage, peripheral cannulation site bleeding, mediastinal cannulation site bleeding, surgical site bleeding | through study completion, an average of 2 years
  Safety and effectiveness outcome
Venous and arterial thromboembolic events | through study completion, an average of 2 years
  Safety and effectiveness outcome
New onset renal replacement therapy (RRT) during ECMO | through study completion, an average of 2 years
  Safety and effectiveness outcome
ECMO free days at day 60 | 60 days
  Safety and effectiveness outcome
ICU free days at day 60 | 60 days
  Safety and effectiveness outcome
Patient Reported Outcome Measure - WHODAS 2.0 | 6 months
  Disability Safety and effectiveness outcome
Patient Reported Outcome Measure - IADL | 6 months
  Independent Activities of Daily Living Safety and effectiveness outcome
Patient Reported Outcome Measure - ADL | 6 months
  Activity of Daily Living Safety and effectiveness outcome
Patient Reported Outcome Measure - MoCA BLIND | 6 months
  Cognitive Function Safety and effectiveness outcome
Patient Reported Outcome Measure - EQ-5D-5L | 6 months
  Quality of Life Safety and effectiveness outcome
Patient Reported Outcome Measure - mRS | 6 months
  Degree of Disability Safety and effectiveness outcome

CONTACTS AND LOCATIONS:
Overall Officials: Hergen Buscher, MBBS, Principal Investigator — St Vincent's Hospital, Sydney; Zoe McQuilten, PhD, Principal Investigator — Monash University; Carol Hodgson, PhD, Principal Investigator — Monash University; Alistair Nichol, PhD, Principal Investigator — Monash University; Aidan Burrell, MBBS, Principal Investigator — Monash University; Mark Dennis, MBBS, Principal Investigator — Royal Prince Alfred Hospital, Sydney, Australia; Timothy Southwood, MBBS, Principal Investigator — Royal Prince Alfred Hospital, Sydney, Australia; Alisa Higgins, PhD, Principal Investigator — Monash University; Sally Newman, Nursing, Principal Investigator — St Vincent's Hospital, Sydney; Thao Le, PhD, Principal Investigator — Monash University
Locations (2):
- Australia (2):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - St Vincent's Health Sydney, Sydney, New South Wales

IPD SHARING:
Plan to Share IPD: No
Patient data is de-identified and only aggregate summaries published.